CLINICAL TRIAL: NCT00676364
Title: A Randomized, Placebo-Controlled Trial to Evaluate Pain and Anxiety During Venipuncture in Pediatric Patients With or Without Pre-treatment by a Topical Anesthetic
Brief Title: Randomized Control Trial of a Topical Anesthetic to Evaluate Pain and Anxiety During Venipuncture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jenny Boucher, PharmD (Other)
Responsible Party: Sponsor-Investigator, Jenny Boucher, PharmD, Investigator, Lehigh Valley Hospital
Organization: Lehigh Valley Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-20030313
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-08

CONDITIONS: Pain; Anxiety
Keywords: pediatric patients; pain; anxiety; topical anesthetic; randomized control trial
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4% lidocaine topical anesthetic cream (Active Comparator): This group received topical 4% lidocaine anesthetic cream under occlusive dressing for 15 minutes prior to needle stick.
  Interventions: Drug: 4% lidocaine topical anesthetic cream
- Placebo (Placebo Comparator): This group received matching placebo cream under occlusive dressing for 15 minutes prior to needle stick.
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: 4% lidocaine topical anesthetic cream — A dollop of 4% lidocaine cream was applied under occlusive dressing for 15 mins prior to venipuncture
  Other Names: 4% liposomal lidocaine (Brand name = LMX4)
  Arms: 4% lidocaine topical anesthetic cream
Drug: Placebo cream — A dollop of matching placebo cream was applied under occlusive dressing for 15 mins prior to venipuncture
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the amount of anxiety and pain felt by children during procedures that require a needle stick after using a topical anesthetic or placebo cream.

DETAILED DESCRIPTION:
Pediatric patients frequently receive eutectic mixture of local anesthetics (EMLA) or other anesthetic medications prior to venipuncture. However, the time for the anesthetic to take affect is approximately 60 minutes. Another anesthetic medication besides EMLA is lidocaine 4% topical anesthetic cream (LMX4), which has a shorter acting time (30 minutes) compared to the EMLA, making it a more desirable medication when urgent labs are required. This medication is being evaluated to assess the anxiety and pain associated with venipuncture in 15 minutes versus the approved 30 minutes of pediatric patients treated as an inpatient or outpatient in the local Emergency Department, compared to standard care (no prior treatment).

ELIGIBILITY:
Inclusion Criteria:

* children ages 5-18 years of age
* treated as an inpatient or outpatient at Lehigh Valley Hospital within the past 24 hours
* venipuncture order, and that order is their initial venipuncture order (required within 30 mins)

Exclusion Criteria:

* known allergy to EMLA, LMX4 or any of their ingredients
* known sensitivities to local anesthetics of the amide type, lidocaine or prilocaine
* G6PD deficiency
* methemoglobinemia or concomitant administration of methemoglobin-inducing agent
* brain injured or disoriented (Glasgow Coma Scale <15)
* cognitively impaired (Mini Mental Status Exam <28)
* active skin conditions at venipuncture site including frequent rashes, eczema or unexplained bruising

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2003-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Boucher, PharmD, Principal Investigator — Lehigh Valley Hospital; Scott Brenner, MD, Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Hospital, Allentown, Pennsylvania, United States

REFERENCES:
- [Background] Koh JL, Fanurik D, Stoner PD, Schmitz ML, VonLanthen M. Efficacy of parental application of eutectic mixture of local anesthetics for intravenous insertion. Pediatrics. 1999 Jun;103(6):e79. doi: 10.1542/peds.103.6.e79. PMID 10353976
- [Background] Lander J, Hodgins M, Nazarali S, McTavish J, Ouellette J, Friesen E. Determinants of success and failure of EMLA. Pain. 1996 Jan;64(1):89-97. doi: 10.1016/0304-3959(95)00100-X. PMID 8867250
- [Background] Eichenfield LF, Funk A, Fallon-Friedlander S, Cunningham BB. A clinical study to evaluate the efficacy of ELA-Max (4% liposomal lidocaine) as compared with eutectic mixture of local anesthetics cream for pain reduction of venipuncture in children. Pediatrics. 2002 Jun;109(6):1093-9. doi: 10.1542/peds.109.6.1093. PMID 12042548
- [Background] Zempsky WT, Cravero JP; American Academy of Pediatrics Committee on Pediatric Emergency Medicine and Section on Anesthesiology and Pain Medicine. Relief of pain and anxiety in pediatric patients in emergency medical systems. Pediatrics. 2004 Nov;114(5):1348-56. doi: 10.1542/peds.2004-1752. PMID 15520120
- [Background] Lander J, Fowler-Kerry S, Oberle S. Children's venipuncture pain: influence of technical factors. J Pain Symptom Manage. 1992 Aug;7(6):343-9. doi: 10.1016/0885-3924(92)90087-x. PMID 1517650
- [Background] Barnett P. Alternatives to sedation for painful procedures. Pediatr Emerg Care. 2009 Jun;25(6):415-9; quiz 420-2. doi: 10.1097/PEC.0b013e3181a93ff3. PMID 19528768
- [Background] Koh JL, Harrison D, Myers R, Dembinski R, Turner H, McGraw T. A randomized, double-blind comparison study of EMLA and ELA-Max for topical anesthesia in children undergoing intravenous insertion. Paediatr Anaesth. 2004 Dec;14(12):977-82. doi: 10.1111/j.1460-9592.2004.01381.x. PMID 15601345
- [Background] Bringuier S, Dadure C, Raux O, Dubois A, Picot MC, Capdevila X. The perioperative validity of the visual analog anxiety scale in children: a discriminant and useful instrument in routine clinical practice to optimize postoperative pain management. Anesth Analg. 2009 Sep;109(3):737-44. doi: 10.1213/ane.0b013e3181af00e4. PMID 19690240
- [Background] Garra G, Singer AJ, Taira BR, Chohan J, Cardoz H, Chisena E, Thode HC Jr. Validation of the Wong-Baker FACES Pain Rating Scale in pediatric emergency department patients. Acad Emerg Med. 2010 Jan;17(1):50-4. doi: 10.1111/j.1553-2712.2009.00620.x. Epub 2009 Dec 9. PMID 20003121
- [Background] Gift AG. Visual analogue scales: measurement of subjective phenomena. Nurs Res. 1989 Sep-Oct;38(5):286-8. No abstract available. PMID 2678015
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Kaweski S; Plastic Surgery Educational Foundation Technology Assessment Committee. Topical anesthetic creams. Plast Reconstr Surg. 2008 Jun;121(6):2161-2165. doi: 10.1097/PRS.0b013e318170a7a4. PMID 18520909

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one site of a multi-site, academic, community emergency department. Children between the ages of five and 18 years of age were considered for enrollment into the study if they were seen in the emergency department (ED) and a physician order was placed for intravenous cannulation or labs to be drawn by venipuncture.
Pre-assignment Details: A convenience sample was utilized due to the availability of the research study coordinator who completed the enrollment from 7 am to 5 pm Monday through Friday. One participant was excluded from analysis due to ineligibility.
Groups:
- ControI Group Receiving Placebo Cream: Control group receiving blinded placebo cream under occlusive dressing prior to venipuncture
- Investigational Group Receiving 4% Lidocaine: Investigational group receiving blinded 4% lidocaine cream under occlusive dressing for 15 mins prior to venipuncture
Period: Overall Study
Arm/Group | ControI Group Receiving Placebo Cream | Investigational Group Receiving 4% Lidocaine
Started | 57 | 57
Completed | 57 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ControI Group Receiving Placebo Cream Before Venipuncture: Experimential group receiving medicated topical cream prior to venipuncture
- Investigational Group: Investigational group receiving blinded 4% lidocaine cream
- Total: Total of all reporting groups
Arm/Group | ControI Group Receiving Placebo Cream Before Venipuncture | Investigational Group | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57 | 57 | 114
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 11.6 (3.7) | 11.6 (3.7) | 11.6 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  United States | 57 | 57 | 114

OUTCOME MEASURES:

1. Secondary Outcome: Anxiety of Venipuncture
Description: Participant anxiety was measured by the study participant and the objective observer before (anticipatory), during (venipuncture) and after (recovery) venipuncture using a validated visual analog scale (VAS). The VAS is a validated scale that is used to detect small changes in many types of observations. The scale ranges from 0-100 scores on a scale, and here the higher scores indicate higher anxiety levels. Only the participant's mean venipuncture (during venipuncture) anxiety scores are presented in outcome measure results here.
Time Frame: During venipuncture
Population: We determined that we will need to enroll 43 children in each group, for a power of .80, alpha=0.05. We used a per protocol analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- ControI Group Receiving Placebo Cream: Control group receiving placebo topical cream prior to venipuncture
- Investigational Group: Investigational group receiving 4% lidocaine cream prior to venipuncture
Arm/Group | ControI Group Receiving Placebo Cream | Investigational Group
Number analyzed (Participants) | 57 | 57
scores on a scale | 43.1 (36.5) | 40.5 (36.4)

2. Primary Outcome: Pain From Venipuncture
Description: Pain was measured immediately after venipuncture by the participant using the six-point FACES scale. "FACES" in not an acronym, but rather a description of a pain scale that uses pictures of faces in various states of pain. The FACES pain scale is a common scale used to measure pain with scores on a scale. The scale we used had six points from zero (0) to five (5) indicating different levels of pain. Lower scores indicate lower levels of pain, and higher scores indicate higher levels of pain.
Time Frame: Pain was measured immediately after venipuncture.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- ControI Group Receiving Placebo Cream: The control group received blinded placebo cream under occlusive dressing for 15 minutes prior to venipuncture.
- Investigational Group Receiving 4% Lidocaine Cream: The investigational group received blinded 4% lidocaine cream under occlusive dressing for 15 minutes prior to venipuncture.
Arm/Group | ControI Group Receiving Placebo Cream | Investigational Group Receiving 4% Lidocaine Cream
Number analyzed (Participants) | 57 | 57
scores on a scale | 2.2 (1.4) | 2.1 (1.6)
Statistical Analysis 1: Comparison: ControI Group Receiving Placebo Cream vs Investigational Group Receiving 4% Lidocaine Cream; P-value determined from linear regression models that include age, gender, number of needle sticks in previous 2 years and nurse reported difficulty in performing venipuncture; Test type: Non-Inferiority or Equivalence — We determined that we will need to enroll 43 children in each group, for a power of .80, alpha=0.05. We used a per protocol analysis; p = 0.71, Chi-squared; Mean Difference (Final Values) = 2.1 — To assess the association between pain and anxiety with intervention group while controlling for other factors, linear regression was used

ADVERSE EVENTS:
Time Frame: The participants were followed for the duration of the study period, an average of three hours.
Arm/Group | ControI Group Receiving Placebo Cream | Investigational Group
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

LIMITATIONS AND CAVEATS:
Convenience sample at one hospital site during dayshift hours Monday through Friday. Variable ages may increase the variance among pain measurements. Analyzed IV cannulation and lab draw together. We did not conduct interrater reliability testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes